CLINICAL TRIAL: NCT01025089
Title: A Phase II Trial of Chemotherapy Plus Cetuximab Followed by Surgical Resection in Patients With Locally Advanced or Recurrent Thymoma or Thymic Carcinoma (BMS #CA225-331/Lilly Trial Alias I4E-US-X007)
Brief Title: Chemotherapy Plus Cetuximab Followed by Surgical Resection in Patients With Locally Advanced or Recurrent Thymoma or Thymic Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry); M.D. Anderson Cancer Center (Other); City of Hope National Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-038
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Thymoma; Thymic Carcinoma; Clinical Masaoka Stage II to IVA
Keywords: Cetuximab; Cisplatin; Cyclophosphamide; 09-038
MeSH Terms: conditions — Thymoma | interventions — Cetuximab; Cisplatin; Doxorubicin; Cyclophosphamide

ARMS (1):
- Cetuximab, Cisplatin, Doxorubicin & Cyclophosphamide (Experimental): This is a multicenter, open-label phase II trial of neoadjuvant chemotherapy and concurrent cetuximab in patients with clinical Masaoka stage II-IVA thymoma or thymic carcinoma.. Patients will initially receive weekly cetuximab for 4 weeks to assess tumor response to cetuximab alone. Patients will then undergo weekly cetuximab along with concurrent CAP for 4 cycles. At the completion of this regimen, patients will undergo surgical resection and the specimen will be evaluated for CPR.
  Interventions: Drug: Cetuximab, Cisplatin, Doxorubicin & Cyclophosphamide

INTERVENTIONS:
Drug: Cetuximab, Cisplatin, Doxorubicin & Cyclophosphamide — Patients will receive single agent cetuximab infusion starting with a 400mg/m2 IV loading dose on day 1 of week 1, followed by weekly infusions (250mg/m2) on day 1 of weeks 2 3, and 4. Patients will receive single agent cetuximab infusion starting with a 400mg/m2 IV loading dose on day 1 of week 1, followed by weekly infusions (250mg/m2) on day 1 of weeks 2 3, and 4. Patients who have completed the neo-adjuvant treatment regimen, who have no evidence of distant progression, and who are medically operable will proceed to surgical resection within 6 weeks of the last infusion.

SUMMARY:
The main purpose of this study is to find out the good and the bad effects that the combination of cetuximab with the traditional chemotherapy regimen of cisplatin, doxorubicin, and cyclophosphamide has when given to patients with later stage thymoma or thymic carcinoma before surgery. The physicians will also look at changes in genes in the tumor that may relate to the effectiveness of cetuximab

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Karnofsky Performance Status (KPS) ≥ 70
* Newly diagnosed or recurrent thymoma - WHO A, AB, B1, B2, or B340, or thymic carcinoma pathologically confirmed at MSKCC, MDACC or City of Hope
* No prior chemotherapy, radiotherapy, or surgical therapy (other than for diagnostic biopsy) for thymoma
* No prior treatment with cetuximab
* Clinical Masaoka Stage II (>5cm), III, or IVA(See Appendix B), including suspected invasion of mediastinum, pericardium, lung, great vessels or chest wall, and/or pleural metastases Normal marrow function: leukocytes ≥ 4,000/μl, absolute neutrophil count ≥ 1,500/μl, platelets ≥ 160,000/μl
* Adequate renal function, with creatinine ≤ 1.3 mg/dl or calculated creatinine clearance ≥60ml/min by Cockcroft and Gault equation using parameters of age, weight (kg), and baseline serum creatinine (mg/dl)
* Adequate hepatic function: Total bilirubin ≤1.5 mg/dl, AST ≤1.5X UNL, alkaline phosphatase ≤1.5 UN
* Signed informed consent
* Effective contraception
* Medically operable

Exclusion Criteria:

* Evidence of distant metastatic disease (Masaoka stage IVB)
* Thymic carcinoid
* Patients must not be receiving any other investigational agents
* Concurrent or prior malignancy in the last 5 years other than non-melanoma skin cancer and in-situ carcinoma of the cervix
* Known HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with the study drugs. Patients on medications known to alter CYP3A4
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the frequency of complete pathologic response to neo-adjuvant therapy with cisplatin, doxorubicin, cyclophosphamide (CAP) and cetuximab in patients with clinical Masaoka stage II-IVa thymoma and thymic carcinomas. | 2 years

SECONDARY OUTCOMES:
To determine the toxicity (CTCAE v.3) of neo-adjuvant therapy with CAP and cetuximab | 2 years
To measure the radiographic response rate to cetuximab alone after 4 weeks | 4 weeks
To determine the radiographic response rate to CAP and cetuximab | 2 years
To determine the complete resection rate (R0) after neo-adjuvant therapy with CAP and cetuximab | 2 years
To correlate percentage of pathologic response to unidimensional and volumetric radiographic response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Huang, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - City of Hope Medical Center, Duarte, California
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm